CLINICAL TRIAL: NCT00227500
Title: A Randomised, Double-Blind Study of Pravastatin for the Treatment of Hyperlipidaemia in Patients With HIV
Brief Title: Pravastatin for Hyperlipidaemia in HIV.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Garvan Institute of Medical Research (Other); St Vincent's Hospital, Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRAVA; PRAVA / RO1 HL65953-01
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2006-06

CONDITIONS: HIV Infections; Lipid Metabolism; Glucose Metabolism; Metabolic Abnormality; Lipodystrophy; Cardiovascular Disease
Keywords: Hyperlipidaemia; Lipid metabolism; Glucose metabolism; HMG CoA reductase inhibitors; Lipodystrophy; Cardiovascular disease; Treatment Experienced; HIV
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Cardiovascular Diseases; Hyperlipidemias | interventions — Pravastatin

INTERVENTIONS:
Drug: Pravastatin

SUMMARY:
This study is a randomised, placebo-controlled study of the effect of treatment with the HMG-CoA reductase inhibitor, pravastatin, in HIV-infected, protease inhibitor treated patients with high serum cholesterol. We hypothesise that pravastatin will result in greater reductions in cholesterol than placebo when used in conjunction with appropriate dietary advice.

DETAILED DESCRIPTION:
High serum cholesterol concentrations are commonly seen in HIV-infected patients treated with some protease inhibitor medications as part of long-term antiretroviral therapy for HIV. There is concern that these elevations in cholesterol may negatively impact on long-term risk of cardiovascular disease in this patient population. Pravastatin, a HMG-CoA reductase inhibitor, is commonly used to treat hypercholesterolaemia in the general population. We aim to examine the effect of 12 weeks therapy with 40mg pravastatin daily in conjunction with dietary advice in HIV-infected patients with elevated serum cholesterol on continued protease inhibitor therapy.

After 4 weeks of dietary advice, patients will be randomised to receive either pravastatin or placebo for 12 weeks. Assessments include fasting lipid and glycaemic parameters, measures of body composition and HIV disease, and surrogate markers for cardiovascular disease.

Although previous small studies of pravastatin in this field have been performed, none has done so in a randomised placebo controlled trial taking into account all the relevant measures.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the trial
* HIV-1 sero-positive
* Male/female >18 years age
* Currently receiving HIV protease inhibitor therapy for > 12 weeks and unlikely to require change in existing regimen during the 16 week study period
* Fasting cholesterol > 6.5 mmol/L (mean of 2 samples collected > 3 days apart)

Exclusion Criteria:

* Any condition which may interfere with ability to comply with study
* Gastrointestinal disorder which may affect drug absorption
* Hypertension or congestive cardiac failure
* Lactic acidemia (serum lactate level >2.2 mmol/L)
* Any serious medical condition which may compromise the patient's safety, including pancreatitis or hepatitis within past 6 months
* Active AIDS defining conditions
* Concurrent therapy with any other lipid lowering agents, oral hypoglycaemics, anabolic steroids or insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-07; Study Completion 2004-10

PRIMARY OUTCOMES:
Between-group difference in time weighted change from baseline in fasting serum total cholesterol

SECONDARY OUTCOMES:
Includes: between-group difference in time weighted change: from wk 4 in fasting serum total cholesterol as well as from baseline in HDL-cholesterol and triglycerides; in total and regional body fat; in endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Carr, MD, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.; David A Cooper, MD, Study Director — National Centre in HIV Epidemiology and Clinical Research.
Locations (1):
- St. Vincents Hospital, Sydney, New South Wales, Australia

REFERENCES:
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/